CLINICAL TRIAL: NCT01649531
Title: Two Implants Versus One Implant With a Cantilever - a Randomized Controlled Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0097
Record Dates: First submitted 2012-07-20; First posted 2012-07-25 (Estimated); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Dental Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test group (Active Comparator): 1 Implant, to be placed in the position with greater vertical bone height with a mesial or distal cantilever.
  Interventions: Procedure: 1 Implant
- Control group (Active Comparator): 2 Implants
  Interventions: Procedure: 2 Implants

INTERVENTIONS:
Procedure: 1 Implant
  Arms: Test group
Procedure: 2 Implants
  Arms: Control group

SUMMARY:
The aim of the present study is to test whether there is a difference in the marginal bone level change between implants with and without cantilevers.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients 18 years to 80 years of age
* no general medical condition which represents a contraindication to implant treatment
* two adjacent missing teeth in the maxilla or mandible in positions of premolars and molars
* at least one tooth present adjacent to the edentulous space
* indication for implant treatment is given
* at least 8 mm of vertical bone height in the mandible allowing for the placement of a 6 mm implant (2 mm safety distance to inferior alveolar nerve)
* at least 4 mm of vertical bone height in the maxilla
* signed informed consent after being informed

Exclusion Criteria:

* smoking of more than 15 cigarettes a day (clinical studies show an increased failure rate of implants in heavy smokers)
* poor oral hygiene after hygienic phase (Plaque Index over 30 %)
* active periodontal disease
* pregnancy or breastfeeding at date of inclusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-08-09 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
radiographic bone level | 5 years
  The primary endpoint of the study is the radiographic bone level 5 years after insertion.The bone level represents an indicator of the osseointegration and biological success of the implant.

SECONDARY OUTCOMES:
Radiographic bone level | 1, 3, 7, 10 years
Implant survival and success | 1, 3, 5, 7, 10 years
rate of technical complication | 1, 3, 5, 7, 10 years
  technical complications: screw loosenings, screw fractures, framework fractures, veneering ceramic fractures
rate of biological complications | 1, 3, 5, 7, 10 years
  biological complications: mucositis, assessed by bleeding on probing
Soft tissue changes | 1, 3, 5, 7, 10 years
  Soft tissue changes: change in clinical crown length = recession / papilla index
Patient morbidity | 1, 3, 5, 7, 10 years
  VAS scale to assess pain after implant placement

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Thoma, Prof. Dr., Principal Investigator — Clinic of Reconstructive Dentistry
Locations (1):
- Center of Dental Medicine Clinic of Reconstructive Dentistry, Zurich, Switzerland

REFERENCES:
- [Derived] Strauss FJ, Schiavon L, Naenni N, Kraus RD, Saenz-Ravello G, Muller N, Jung RE, Thoma DS. Cost Effectiveness of Two Short Implants Versus One Short Implant With a Cantilever in the Posterior Region: 7.5-Year Follow-Up of a Randomised Controlled Trial. J Clin Periodontol. 2025 Dec;52(12):1712-1724. doi: 10.1111/jcpe.70039. Epub 2025 Sep 21. PMID 40976576
- [Derived] Thoma DS, Wolleb K, Schellenberg R, Strauss FJ, Hammerle CHF, Jung RE. Two short implants versus one short implant with a cantilever: 5-Year results of a randomized clinical trial. J Clin Periodontol. 2021 Nov;48(11):1480-1490. doi: 10.1111/jcpe.13541. Epub 2021 Sep 22. PMID 34448219